CLINICAL TRIAL: NCT03025399
Title: Multi Center Clinical Study of Chinese Medicine Intervention on Early Diabetic Microvascular Complications: Multi Centers Clinical Study of Tang Wang Prescription Intervene Diabetic Non-proliferative Retinopathy
Brief Title: Clinical Study of Tang Wang Prescription Intervene Diabetic Non-proliferative Retinopathy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fengmei Lian (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Zhengzhou City Hospital of Traditional Chinese Medicine (Other); Baodin City Hospital of Traditional Chinese Medicine (Unknown); zi bo wanjie cancer hospital (Unknown); Shijiazhuang City Hospital of Traditional Chinese Medicine (Unknown); Zouping Country Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Fengmei Lian, Chief, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015Tangwang Prescription
Record Dates: First submitted 2017-01-04; First posted 2017-01-19 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetic Non-proliferative Retinopathy; Type2 Diabetes
Keywords: tang wang prescription

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tangwang Prescription (Experimental): The prescription was composed five Chinese herbal medicines,every bag has 4.87g granules, take it one bag each time, two times a day.
  Interventions: Drug: Tangwang prescription
- Placebo (Placebo Comparator): Placebo is a simulated drug of tangwang Prescription,every bag has 4.87g granules, take it one bag each time, two times a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tangwang prescription — A kind of Granule(Tangwang prescription) was composition by five Chinese herbal medicines, every bag has 4.87g granules.
  Other Names: Tang Wang Fang
  Arms: Tangwang Prescription
Drug: Placebo — Placebo is a simulated drug of tangwang prescription,included weight, appearance, colour, taste,smell and solubility.
  Other Names: Placebos
  Arms: Placebo

SUMMARY:
This study include 384 Participants with diabetic non-proliferative retinopathy

Design Method: Randomized, double blind, placebo controlled and multicenter clinical study. Participants treatment for 48 weeks, and main aimed to evaluate the therapeutic effect of tang wang prescription improve degree of retinal microvascular disease of patients with diabetic non-proliferative retinopathy.

DETAILED DESCRIPTION:
1. This study is a randomized, double-blinded, placebo-controlled and multicenter clinical trial on type 2 diabetic non-proliferative retinopathy to evaluate the therapeutic effect of tang wang prescription.
2. Through the calculation of sample size, 384 participants with type 2 diabetic non-proliferative retinopathy will be recruited for the study, all participants were randomly divided into 2 groups, and both of groups would be performed on a basic treatment (including diabetes education, diabetes diet, rational control of blood glucose (oral hypoglycemic agents or insulin injections to keep all participants keep blood glucose stable in the study. If fasting blood glucose fluctuates more than 20%, need to find and remove the factors as soon as possible, and adjust the dose and monitor change of blood glucose, make it smooth in 4 weeks. Adjusted dose of the drug needs to be detailed records in the combined medication table), and oral calcium dobesilate treatment), study group take tang wang prescription, take one bag each time and twice on day, control group take the same dose of placebo.
3. The study will last for 48 weeks. Once every four weeks follow-up, color fundus photography, fundus fluorescein angiography, and coherent optical tomography were performed every six months; ETDRS international visual acuity test was performed every months.
4. Curative effect evaluation criteria:

   * Main evaluation criteria: the changes of degree of retinal microvascular lesions before and after treatment, according to the change of degree of retinal microvascular lesions (no, mild non proliferative phase, moderate non proliferative phase, severe non proliferative phase, proliferative phase), divided into aggravated, unchanged, reduce three conditions. Aggravated was defined as the degree of retinal microvascular lesions severity more than grade 1 after treatment; unchanged was defined as the degree of retinal microvascular lesions before and after treatment did not change; reduce was defined as the degree of retinal microvascular lesions reduced more than 1 grade after treatment.
   * Second evaluation criteria:

     * Change of the number of micro hemangioma of diabetic retinopathy before and after treatment;
     * Change of the number of microvascular bleeding of diabetic retinopathy before and after treatment;
     * Change of the number of microvascular leakage of diabetic retinopathy before and after treatment;
     * Degree of change of macular edema of diabetic retinopathy before and after treatment;
     * Change of Vision before and after treatment.
5. Diagnostic and monitoring indicators：blood pressure, fasting blood glucose test (every one month); glycated hemoglobin, blood lipids (every three months); Routine eye examination and fundus examination, including intraocular pressure, anterior segment, lens, vitreous body, and lens, vitreous need describe the conditions of opacity (every six months).
6. The provisions of the combined therapy

   * All Chinese herbal medicines with the same efficacy as the study drug (including Chinese herbal medicines with similar therapeutic and similar efficacy in Instructions) were banned during the study period.
   * All combined therapy and Combined medication(treatment measure or treatment medicine of other diseases) should be recorded in the combined medication table.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diabetic retinopathy、the degree of disease was non-proliferative diabetic retinopathy；
2. Age at 30-70 years old；
3. Signed the informed consent；

   * Note: Diabetic retinopathy patients can be selected as the observation object, Who only one eye can meet the inclusion criteria, If both eyes of patient can be selected, please record respectively, and choose one eye to evaluate the curative effect, the eye must according to the following principles: choose the heavier eye as the observation eye, When the fundus conditions of the eyes are in different clinical stages; Select the eye as the eye of clinical manipulation. Choose the eyes with better clinical operation as the observation eyes, When the fundus conditions of the eyes are in same clinical stages.

Exclusion Criteria:

1. The patients with retinal photocoagulation、appropriate patients for retinal photocoagulation、patient have one or two eyes in diabetic retinopathy proliferative phase、type I diabetes mellitus、there are other eye disease complications(such as glaucoma、cataracts can Significantly interfere the fundus examination、Non - diabetic retinopathy、uveitis、amotio retinae、optic nerve diseases and high myopia with fundus lesions et al.)
2. Combined with severe primary disease such as cardiovascular、liver、kidney and hematopoietic system et al、the serum transaminase was 2 times larger than the normal valuet、Serum creatinine greater than the upper limit of normal value、Psychiatric patients.
3. Women with Pregnancy or prepare for pregnancy or lactating.
4. Patient participated in other clinical researchers within a month.
5. Patients have been treated with other drugs to treat diabetic retinopathy except for calcium hydroxide within a week.
6. Systolic blood pressure > 160mmHg or diastolic blood pressure > 100mmHg.
7. Patients with diabetic ketosis, ketoacidosis and severe infections within a month
8. Patients have been alcohol abused and / or used psychoactive substances or drug abused or drug addicted within 5 years.
9. According to the researcher's judgment, patients have Other lesions or conditions maybe reduce the possibility of entering groups or make the groups complex,such as working environment change frequently、Living environment is unstable what easy to cause loss to follow-up.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
the changes of degree of retinal microvascular lesions before and after treatment (no, mild non proliferative phase, moderate non proliferative phase, severe non proliferative phase, proliferative phase) | 0 week, 24 weeks, 48 weeks

SECONDARY OUTCOMES:
Change of the number of micro hemangioma of diabetic retinopathy | 0 week, 24 weeks, 48 weeks
Change of the number of microvascular bleeding of diabetic retinopathy | 0 week, 24 weeks, 48 weeks
  Color fundus photography and fundus fluorescein angiography were performed
Change of the number of microvascular leakage of diabetic retinopathy | 0 week, 24 weeks, 48 weeks
Degree of change of macular edema of diabetic retinopathy,analysis of measured values of the shortest distance from the margin of edema and the retinal thickness in macular region before and after medication | 0 week, 24 weeks, 48 weeks
Change of Vision (analysis of visual acuity before and after medication using EDTRS international visual acuity chart) | 0 week, 4 weeks, 8 weeks,12 weeks,16 weeks, 20 weeks, 24 weeks, 28 weeks, 32 weeks, 36 weeks, 40 weeks, 44 weeks, 48 weeks

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jin D, Zhang Y, Zhang Y, Huang W, Meng X, Yang F, Bao Q, Zhang M, Yang Y, Ni Q, Lian F, Tong X. Efficacy and Safety of TangWang Prescription for Type 2 Non-Proliferative Diabetic Retinopathy: A Study Protocol for a Randomized Controlled Trial. Front Pharmacol. 2021 Mar 15;12:594308. doi: 10.3389/fphar.2021.594308. eCollection 2021. PMID 33790783